CLINICAL TRIAL: NCT05843604
Title: Cerebral and Cognitive Markers of Treatment Resistance in Obsessive-compulsive Disorder: Towards Personalization of Patient Care
Brief Title: Cerebral and Cognitive Markers of Treatment Resistance in Obsessive Compulsive Disorder
Acronym: 3TOC
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00463-40
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: OCD
Keywords: functional MRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obsessive compulsive disorder patients
  Interventions: Other: Functional MRI
- Control Patients
  Interventions: Other: Functional MRI

INTERVENTIONS:
Other: Functional MRI — Three cognitive tests will be performed in the MRI, namely a stroop task, an N-back task and a switching task

SUMMARY:
This study aims to define individual profiles of treatment resistants in order to find indicators and predictors of the therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Obsessive compulsive disorder diagnosed according to Diagnostic and Statistical Manual 5 criteria (patients will be included regardless of the severity and resistance of their pathology and their levels of executive functions)
* Understand and accept the constraints of the study
* Be a beneficiary or affiliated to a Health Insurance scheme

Exclusion Criteria:

* Present one of the diagnoses according to the criteria of the DSM 5: schizophrenic disorders, substance abuse or dependence to a substance according to the criteria of the M.I.N.I. version 5.0 (Sheehan et al., 1998)
* Generalized anxiety disorder, social anxiety, nicotine dependence and history of a major depressive episode are not exclusion criteria according to the M.I.N.I. version 5.0 (Sheehan et al., 1998)
* Have a serious intercurrent pathology
* Being a pregnant woman
* Being a woman of childbearing age without effective contraception.
* Being hospitalized under duress or on an outpatient basis in a care program
* Being under judicial protection (reinforced curatorship, guardianship)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Clinical Research Unit of Poitiers. All volunteer patients included in this study will be included regardless of the degree of resistance to treatment or the severity of their disease. Patients will not be hospitalized for the duration of the study unless their condition requires it.
  Healthy volunteers will be recruited locally by advertisement or through acquaintances, and will be matched to each patient based on age, gender, laterality, and education level. They must not have an acute pathology being treated, nor take psychotropic drugs, nor be followed in psychotherapy. In their history, we must not find hospitalization in a psychiatric environment or a psychiatric illness according to the M.I.N.I. version 5.0.0.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Cerebral activity modification during N-back task | Day 1
  Blood-oxygen-level-dependent (BOLD) modification during the task between obsessive compulsive disorder patients and controls
Cerebral activity modification during Stroop task | Day 1
  Blood-oxygen-level-dependent (BOLD) modification during the task between obsessive compulsive disorder patients and controls
Cerebral activity modification during switching task (Monsell et Mizon task ) | Day 1
  Blood-oxygen-level-dependent (BOLD) modification during the task between obsessive compulsive disorder patients and controls

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided